CLINICAL TRIAL: NCT01806090
Title: Uninterrupted Clopidogrel Therapy Before Elective Colonoscopy Will Increase the Risk of Post-polypectomy Bleeding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Francis KL Chan, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCP
Record Dates: First submitted 2013-03-04; First posted 2013-03-07 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Gastrointestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clopidogrel (Active Comparator): Continue clopidogrel for 7 days prior to the endoscopic procedure
  Interventions: Drug: clopidogrel
- Placebo (Placebo Comparator): Placebo daily for 7 days prior to the endoscopic procedure
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: clopidogrel — Clopidogrel 7 days prior to the endoscopic procedure (Colonoscopy)
  Other Names: Plavix
  Arms: Clopidogrel
Other: Placebo — Placebo for 7 days prior to the endoscopic procedure (Colonoscopy)
  Arms: Placebo

SUMMARY:
This double-blind, randomized trial aims to evaluate whether uninterrupted anti-platelet therapy (clopidogrel) will increase the risk of bleeding associated with removal of polyp during colonoscopy in patients with coronary artery disease.

DETAILED DESCRIPTION:
Clopidogrel is a potent anti-platelet agent that, when combines with aspirin, is essential in treating acute myocardial infarction and preventing coronary stent thrombosis. However, adding clopidogrel to aspirin has been shown to substantially increase the risk of gastrointestinal bleeding by 70%. This increased bleeding risk is a particular concern for patients requiring colonoscopy. The latter is a gold standard for screening colorectal cancer. This endoscopic procedure is increasingly performed for patients on anti-platelet drugs because coronary artery disease is associated with increased risk of colorectal neoplasia. We have shown that over 30% of patients with coronary artery disease have colorectal neoplasia.

Management of patients on clopidogrel who undergo colonoscopy is a clinical dilemma. Continuation of clopidogrel may increase the risk of bleeding associated with endoscopic resection of polyps (post-polypectomy bleeding). This is a potentially serious complication because post-polypectomy bleeding is often delayed, difficult to locate, and may provoke acute coronary syndrome. Conversely, prolonged discontinuation of clopidogrel increases the risk of recurrent myocardial infarction and coronary stent thrombosis.

There is a lack of prospective data on the risk of post-polypectomy bleeding attributable to clopidogrel. Current American Society of Gastrointestinal Endoscopy and British Society of Gastroenterology Guidelines recommend withholding clopidogrel for 7 to 10 days in planned high risk endoscopic procedures such as colonoscopic polypectomy. However, this guideline is largely based on retrospective data and expert opinion. In fact, the anti-platelet effect of clopidogrel lasts for about 5 days only. Coronary stent thrombosis has been reported as early as 7 days after stopping clopidogrel. There remains a large gap in our knowledge on the risk of bleeding in patients taking clopidogrel who undergo gastrointestinal endoscopic procedures.

No randomized trials have assessed whether clopidogrel should be discontinued before colonoscopy. This randomized trial aims to assess whether uninterrupted clopidogrel therapy during colonoscopy will increase the risk of post-polypectomy bleeding. Irrespective of the outcome, this trial will be the first to provide controlled data on the risk of post-polypectomy bleeding with uninterrupted clopidogrel during colonoscopy. Unfortunately, this important clinical question is not a priority of pharmaceutical companies because clopidogrel will be off patent soon. The outcome of this industry-independent clinical trial may encourage health authorities and international guideline committees to review their recommendations on the management of anti-platelet therapy for high-risk endoscopic procedures.

Hypothesis Uninterrupted clopidogrel therapy increases the risk of post-polypectomy bleeding in patients undergoing elective colonoscopy

Aim To investigate whether uninterrupted clopidogrel therapy before elective colonoscopy will increase the risk of post-polypectomy bleeding

Study Design This is a double-blind, randomized, controlled trial in which patients receiving clopidogrel for coronary stents who require elective colonoscopy will be randomized to either clopidogrel or its placebo for one week prior to the endoscopic procedure

Colonoscopic Procedures Experienced colonoscopists will perform colonoscopy under conscious sedation with midazolam and pethidine. Bowel preparation consists of polyethylene glycol taken orally the evening and the morning before procedure together with a minimum of 2 liters of clear fluids. The adequacy of bowel preparation will be documented (poor, fair, good, or excellent). Colonoscopists will be instructed to remove all polyps during the colonoscopic examination. The location and morphologic feature of each polyp will be recorded. The size is measured using an open biopsy forceps (6 mm apart). Each lesion will be fixed in formalin and sent to the pathologist for histologic evaluation. No prophylactic clips or detachable loops will be applied if immediate bleeding is not observed after polypectomy. Intervention for immediate post-polypectomy bleeding including injection therapy alone or in combination with endoclip application, if any, will be recorded.

Follow-up assessment All patients will resume their usual prescriptions of clopidogrel after colonoscopy when oral intake is allowed. They will be monitored hourly for hemodynamic instability and any delayed post-polypectomy bleeding for 24 hours. After discharge, a designated research nurse will contact the patients by telephone on Day 2 and Day 7 for symptoms of bleeding. On Day 30, they will return for a full blood count and symptoms of delayed post-polypectomy bleeding. Emergency visits and hospital discharge summaries will be scanned for up to 6 months after colonoscopy for recurrent cardiothrombotic events. A 24-hour hotline will be provided for patients to report any adverse or serious events.

ELIGIBILITY:
Inclusion Criteria:

1. On regular treatment with clopidogrel alone or in combination with other anti-platelet drugs (e.g. aspirin)
2. Elective colonoscopy for asymptomatic screening of bowel cancer or investigation of bowel symptoms (e.g. altered bowel habit, rectal bleeding, anemia, polyp follow-up)
3. Age ≥ 18
4. Written informed consent

Exclusion Criteria:

1. Coronary stent of any type placed within 30 days
2. Cardiac-vascular event within 3 months
3. Drug-eluting coronary stent placed within 6 months
4. Terminal illness
5. Concomitant use of anticoagulants
6. Congenital or acquired bleeding diathesis showing clinical bleeding tendency (e.g. hemophilia, decompensated cirrhosis)
7. Pregnancy or women of child-bearing age without regular use of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Delayed post-polypectomy bleeding | 30 days post-colonoscopy
  The primary endpoint is delayed post-polypectomy bleeding. The latter is defined as rectal bleeding, starting after the colonoscope has been retracted from the anus to 30 days after the procedure.

SECONDARY OUTCOMES:
Immediate post-polypectomy bleeding | Within 5 minutes after polypectomy
  bleeding at the time of polypectomy that persists despite continuous irrigation with diluted epinephrine solution for 5 minutes.
Serious Cardiothrombotic events | 6 months after colonoscopy
  defined according to the antithrombotic trialists' criteria

CONTACTS AND LOCATIONS:
Overall Officials: Francis KL Chan, MD, Principal Investigator — CUHK
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Chan FKL, Kyaw MH, Hsiang JC, Suen BY, Kee KM, Tse YK, Ching JYL, Cheong PK, Ng D, Lam K, Lo A, Lee V, Ng SC. Risk of Postpolypectomy Bleeding With Uninterrupted Clopidogrel Therapy in an Industry-Independent, Double-Blind, Randomized Trial. Gastroenterology. 2019 Mar;156(4):918-925.e1. doi: 10.1053/j.gastro.2018.10.036. Epub 2018 Oct 25. PMID 30518511